CLINICAL TRIAL: NCT05077449
Title: A Phase III Study to Evaluate the Efficacy and Safety of XZP-3287 in Combination With Fulvestrant Versus Placebo Combined With Fulvestrant in Patients With HR Positive and HER2 Negative Recurrent/Metastatic Breast Cancer
Brief Title: A Study of XZP-3287 in Combination With Fulvestrant in Patients With Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XZP-3287-3001
Record Dates: First submitted 2021-09-18; First posted 2021-10-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Advanced Breast Cancer
Keywords: XZP-3287; HR positive and Her2 negative; recurrent/metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XZP-3287+Fulvestrant (Experimental)
  Interventions: Drug: XZP-3287+Fulvestrant
- Placebo + Fulvestrant (Placebo Comparator)
  Interventions: Drug: Placebo + Fulvestrant

INTERVENTIONS:
Drug: XZP-3287+Fulvestrant — XZP-3287 360 mg orally Twice daily(Q12H) of every 28-day cycle Fulvestrant 500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle (28-day) until progressive disease
  Arms: XZP-3287+Fulvestrant
Drug: Placebo + Fulvestrant — Placebo 360 mg orally Twice daily(Q12H) of every 28-day cycle Fulvestrant 500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle (28-day) until progressive disease
  Arms: Placebo + Fulvestrant

SUMMARY:
This is a phase III clinical trial to evaluate the efficacy and safety of XZP-3287 in combination with Fulvestrant versus placebo combined with Fulvestrant in Patients who have HR positive and Her2 negative recurrent/metastatic breast cancer and have received prior endocrine therapy are eligible for study.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years old;
2. Patient is in the menopausal state；
3. Pathologically-confirmed HR positive and Her2 negative Breast Cancer;
4. Locally advanced stage, recurrence or metastasis breast cancer; 4.1 Disease progression after previous endocrine therapy； 4.2 One previous line of chemotherapy for advanced/metastatic disease is allowed in addition to endocrine therapy;
5. At least one measurable lesion (based on RECIST v1.1) or only bone metastases;
6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
7. Adequate organ and marrow function;
8. Patient of childbearing age must undergo a serum pregnancy test within 14 days before randomization, and the result is negative; patient is willing to use a medically approved high-efficiency contraceptive method during the study period and within 6 months after the last study drug treatment;
9. Patient with acute toxic reactions caused by previous anti-tumor treatments or surgical operations were alleviated to grade 0 to 1 (NCI-CTCAE v5.0), or to the level specified by the enrollment criteria;
10. Patient has signed informed consent before any trial related activities.

Exclusion Criteria:

1. Patient with visceral crisis, inflammatory breast cancer, or brain metastases, except for patient with stable brain metastases;
2. Patient had clinically significant pleural effusions, ascites effusions, or pericardial effusions in the 4 weeks before enrollment;
3. Patient who received prior treatment with mTOR inhibitors, CDK4/6 inhibitors or fulvestrant;
4. Participation in a prior treatment of major surgery, chemotherapy, radiotherapy, and any anti-tumor treatment within 14 days before enrollment；
5. Patient who participated in other clinical trials within 14 days before enrollment or within 5 half-lives of the trial drug, whichever is longer;
6. Patient used CYP3A4 potent inhibitors or potent inducers within 14 days before enrollment or within 5 half-lives of the drug, whichever is longer;
7. Patient who used bisphosphonates or RANKL inhibitors within 7 days before enrollment, patient who have started treatment during the study should not change the method of use;
8. Any other malignant tumor has been diagnosed within 3 years before randomization;
9. Patient is in the active stage of HBV, HCV or co-infected with HBV, HCV, or Patient with positive HIV antibody;
10. Patient with severe infection within 4 weeks before enrollment, or unexplained fever> 38.5℃ during screening/before enrollment;
11. Patient with heart function impaired or clinically significant heart disease within 6 months before enrollment;
12. Cerebrovascular accident occurred within 6 months before enrollment, including history of transient ischemic attack or stroke; symptomatic pulmonary embolism;
13. Inability to swallow, intestinal obstruction or other factors that affect the taking and absorption of the drug;
14. Patient with a known hypersensitivity to any of the excipients in this study;
15. A prior history of autologous or allogeneic hematopoietic stem cell transplantation;
16. A prior history of psychotropic drug abuse or drug use;
17. Pregnant or breastfeeding;
18. The researchers considered that there were some cases that were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression free survival (PFS) | Up to approximately 24 months
  An interim analysis will be performed in this study. The primary endpoint of the study is PFS. An interim analysis is scheduled upon the collection of 70%(approximately 125) PFS events, and the final PFS analysis will be conducted after 178 PFS events have been collected.

SECONDARY OUTCOMES:
BICR-assessed progression free survival (PFS) | Up to approximately 24 months
Overall survival (OS) | Up to approximately 5 years
Overall survival rate(OSR) | Up to approximately 5 years
Objective response rate (ORR) | Up to approximately 24 months
Duration of response (DoR) | Up to approximately 24 months
Disease control rate (DCR) | Up to approximately 24 months
Clinical benefit rate (CBR) | Up to approximately 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to approximately 24 months
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | Up to approximately 24 months
Maximum Plasma Concentration [Cmax] | Up to approximately 4 months
Time to Maximum Plasma Concentration [Tmax] | Up to approximately 4 months
Area under the time-concentration Curve [AUC] | Up to approximately 4 months

OTHER OUTCOMES:
EORTC QLQ-C30 scale | Up to approximately 24 months
EORTC QLQ-BR23 scale | Up to approximately 24 months
EQ-5D-5L scale | Up to approximately 24 months
Plasma ctDNA | Up to approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Science, Beijing, Beijing Municipality, China